CLINICAL TRIAL: NCT05027009
Title: Effects of Simulated Solar Radiation on Human Skin
Brief Title: Effects of Simulated Solar Radiation on Human Skin in Preventing Skin Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Pamela Cassidy, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00022830; NCI-2021-06210 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00022830 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-08-25; First posted 2021-08-30 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (low dose simulated sunlight) (Experimental): Patients undergo total body exam. The minimum dose of simulated sunlight required to cause mild sunburn is determined. One of the patient's moles is exposed to 3 times that minimum dose of simulated sunlight. One day later, that mole, and an untreated mole, are removed by punch biopsy.
  Interventions: Procedure: Physical Examination; Other: Solar Simulated Light
- Group II (middle dose simulated sunlight) (Experimental): Patients undergo total body exam. The minimum dose of simulated sunlight required to cause mild sunburn is determined. One of the patient's moles is exposed to 4 times that minimum dose of simulated sunlight. One day later, that mole, and an untreated mole, are removed by punch biopsy.
  Interventions: Procedure: Physical Examination; Other: Solar Simulated Light
- Group III (high dose simulated sunlight) (Experimental): Patients undergo total body exam. The minimum dose of simulated sunlight required to cause mild sunburn is determined. One of the patient's moles is exposed to 6 times that minimum dose of simulated sunlight. One day later, that mole, and an untreated mole, are removed by punch biopsy.
  Interventions: Procedure: Physical Examination; Other: Solar Simulated Light

INTERVENTIONS:
Procedure: Physical Examination — Undergo total body exam
  Other Names: Assessment; General Examination; Physical; Physical Assessment; Physical Exam; physical_exam
Other: Solar Simulated Light — Undergo exposures to simulated sunlight
  Other Names: Artificial Sunlight; Full-Spectrum Lighting; Solar Simulated Radiation; SSR

SUMMARY:
This clinical trial examines the effects of simulated solar radiation on human skin in preventing skin cancer. Testing whether new drugs affect biomarkers in the skin is a good first test of whether the drug might prevent skin cancer. Some biomarkers in skin, and even in moles, are affected after a person is exposed to sunlight. This study may help doctors learn more about what happens to the skin and moles when the participants are exposed to the sun.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To identify biomarkers of simulated solar radiation (SSR) treatment in human skin that can be used as surrogate endpoints in chemoprevention trials in humans.

SECONDARY OBJECTIVE:

I. Measure Langerhans cell (LC) and sunburn cell density in the epidermis, as well as deoxyribonucleic acid (DNA) damage.

EXPLORATORY OBJECTIVE I. To perform gene expression analysis on tissue frozen after biopsy.

OUTLINE: Patients are randomized to 1 of 3 groups.

GROUP I: Patients undergo total body exam. The minimum dose of simulated sunlight required to cause mild sunburn is determined. One of the patient's moles is exposed to 3 times that minimum dose of simulated sunlight. One day later, that mole, and an untreated mole, are removed by punch biopsy.

GROUP II: Patients undergo total body exam. The minimum dose of simulated sunlight required to cause mild sunburn is determined. One of the patient's moles is exposed to 4 times that minimum dose of simulated sunlight. One day later, that mole, and an untreated mole, are removed by punch biopsy.

GROUP III: Patients undergo total body exam. The minimum dose of simulated sunlight required to cause mild sunburn is determined. One of the patient's moles is exposed to 6 times that minimum dose of simulated sunlight. One day later, that mole, and an untreated mole, are removed by punch biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-100 years. The investigators anticipate recruiting few if any patients over age 80 as nevi tend to disappear as people age. Both men and women of all races and ethnic groups will be included
* Participants must have 2 clinically benign melanocytic nevi 3-5 mm in diameter confirmed by clinical dermatoscopic examination by a medically-qualified study team member and suitable for biopsy (i.e. not at a site that would be functionally or cosmetically damaged by the biopsy). The minimum size restriction arises from the need for collection of tissue sufficient for single nucleus ribonucleic acid sequencing (RNAseq) analysis. The maximum size is dictated by the requirement that the entire nevus be removed with a 6 mm punch biopsy, thereby eliminating any concerns that might arise from regrowth of the nevus that can happen after incomplete removal
* All participants must be able to understand and be willing to sign a written informed consent document

Exclusion Criteria:

* Undergoing systemic therapy for melanoma or any other cancer
* Sensitivity to anesthetic agent
* Photosensitivity
* Currently taking supplements such as nicotinamide or antioxidants that might protect from skin cancer or alter the response of their skin to simulated solar radiation (SSR)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Percentage of pixels positive for p53 by immunohistochemical analysis | Up to 1 year
  Will use immunohistochemical (IHC) analysis of biopsies to determine the difference between the percentage of pixels classified as positive or strong positive for p53 in irradiated nevi (moles) and unirradiated control nevi from each participant. Difference will be measured in percentage points ranging from 0 to 100 with no transformation prior to analysis.

SECONDARY OUTCOMES:
Deoxyribonucleic acid (DNA) damage | Up to 1 year
  Will use IHC analysis of biopsies to examine the difference between the percentage of nuclei in 3 high-powered fields classified as positive or strong positive for cyclobutane pyrimidine dimers (CPDs) or 8-oxoguanine in irradiated nevi and unirradiated control nevi from each participant. Differences will be measured in percentage points ranging from 0 to 100 with no transformation prior to analysis.
Difference in the number of sunburn cells per high power field in irradiated and unirradiated control nevi | Up to 1 year
  Will use immunohistochemical analysis of biopsies to examine the difference between the number of apoptotic keratinocytes (sunburn cells) in irradiated nevi and unirradiated control nevi from each participant. Differences will be measured in percentage points ranging from 0 to 100 with no transformation prior to analysis.
Percent of the area of the epidermis that is positive for Langerhans cells | Up to 1 year
  Will use immunohistochemical analysis of biopsies to examine the difference between the area of the epidermis positive for Cd1a in irradiated and unirradiated control nevi. Differences will be measured in percentage points ranging from 0 to 100 with no transformation prior to analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Cassidy, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States